CLINICAL TRIAL: NCT05492526
Title: Using Body Data for the Purpose of Contextualised Feedback to Enable Established Physical Activity Guidelines to be Delivered in a Free- Living Environment as Part of a Comprehensive Cardiac Rehabilitation Programme.
Brief Title: The Use of Contextualised Body Data in Cardiac Rehabilitation (CR)
Acronym: KiCS1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Collaborators: KiActiv (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 4807
Record Dates: First submitted 2022-07-20; First posted 2022-08-08 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2022-07

CONDITIONS: Cardiac Rehabilitation
Keywords: Cardiac Rehabilitation; Myocardial Infarction; CABG; NSTEMI; STEMI; Angina; Exercise; Physical activity; Heart failure; Digital Health
MeSH Terms: conditions — Myocardial Infarction; Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction; Angina Pectoris; Motor Activity; Heart Failure

STUDY DESIGN:
Intervention Model Description: Prospective, randomised, open -label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Cardiac Rehabilitation (Other): Patients receive usual care and wear Ki monitor - doesn't receive any feedback during the cardiac rehabilitation period.
  Interventions: Device: Ki Monitor without feedback
- Intervention Arm - Usual Cardiac Rehabilitation plus contextualised Data feedback (Experimental): Patient receives usual care and also wears Ki monitor and receives contextualised data feedback
  Interventions: Device: Ki monitor with contextualised data feedback

INTERVENTIONS:
Device: Ki Monitor without feedback — Physical activity Monitor - No feedback
  Arms: Usual Cardiac Rehabilitation
Device: Ki monitor with contextualised data feedback — Physical activity monitor and feedback
  Arms: Intervention Arm - Usual Cardiac Rehabilitation plus contextualised Data feedback

SUMMARY:
KiCS1 study : Digital health for current hospital- based Cardiac rehabilitation programmes to increase effectiveness and patient outcomes.

DETAILED DESCRIPTION:
Cardiac rehabilitation (CR) after a heart attack has shown to be more effective than any other medication given after such an event. It is a recommended therapy by NICE. However, only 44% of eligible patients attend rehabilitation and only half of these complete the course. Novel ways to increase uptake and compliance are needed.

In this study, calorie burn and physical activity data will be collected using a validated, CE marked physical activity monitor, herein referred to as Ki monitor. Data can be uploaded to an online behaviour change platform that incorporates personalised feedback in the context of their bespoke requirements for CR to empower people to self-care at home using their personal everyday physical activity. This can be closely monitored and support can be given on the contextualised feedback by healthcare professionals. A small pilot study has been carried out to establish wearability of a physical activity monitor in a CR cohort, which has demonstrated a high level of acceptability.

We now wish to extend this pilot to a randomised study designed to test the effectiveness of using contextualised body data to influence physical activity in a free-living environment amongst patients undergoing CR, based on the current ACPICR standards for Daily Activity and At-home Training. All patients referred for CR will be invited to take part. These will be randomised to the usual care (UC) group or the contextualised data feedback (CDF) group. Both groups will wear the Ki monitor for eight weeks. The UC group will receive usual care, the CDF group will receive usual care with the addition of contextualised feedback on their activities based on the physical activity data.

ELIGIBILITY:
Inclusion Criteria:

All patients referred to the cardiac rehab programme will be invited to take part in the study.

Exclusion Criteria:

1. Individuals using a pacemaker or other internal medical device.
2. Unable to access a computer or tablet with internet access to view the online platform.
3. Unable to access a smartphone or tablet with bluetooth connectivity and internet access to upload data from the activity monitor.
4. Unwillingness to take part.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Achieving the ACPICR standards for physical activity in a free-living environment objectively measured using the Ki monitor | 6 - 8 weeks
  Objective measurement using Ki monitor.

SECONDARY OUTCOMES:
Exercise test result. | 6-8 weeks
  Incremental shuttle walk test or 6 minute walking test, as appropriate
Total calories burned | 6-8 weeks
  Objectively measured using the Ki monitor
Completion of cardiac rehabilitation programme | 6-8 weeks
  Number of participants completed full cardiac rehabilitation programme.

OTHER OUTCOMES:
Quality of life measured using the Dartmouth Coop | 6-8 weeks
  Participants completed a questionnaire at the start and end of the cardiac rehabilitation program.
Anxiety and depression score measured using Hospital Anxiety and depression scale (HADS) | 6-8 weeks
  Participants completed a questionnaire at the start and end of the cardiac rehabilitation program.
Body mass index measured using height and weight and combined to report in kg/m2 | 6-8 weeks
  Measured at the beginning and end of Cardiac rehabilitation programme
Blood pressure measured and reported in mmHg | 6- 8 weeks
  Measured before and after exercise tests at the beginning and end of the cardiac rehabilitation programme
Blood Glucose measured and reported in mmol/L | 6-8 weeks
  Measured at the beginning and end of Cardiac rehabilitation programme where appropriate

CONTACTS AND LOCATIONS:
Overall Officials: Micheal Fisher, Principal Investigator — Liverpool University Hospitals NHS Trust
Locations (1):
- Liverpool University Hospital NHS Foundation Trust, Liverpool, United Kingdom